CLINICAL TRIAL: NCT04191304
Title: A Multicentre, Randomised, Double-blind, Parallel-group, Placebo-controlled, 24-Week Phase III Study With an Open-label Extension to Evaluate the Efficacy and Safety of Benralizumab in Patients With Hypereosinophilic Syndrome (HES)
Brief Title: A Phase III Study to Evaluate the Efficacy and Safety of Benralizumab in Patients With Hypereosinophilic Syndrome (HES)
Acronym: NATRON
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3254C00001; 2023-510455-28-00 (Registry Identifier: CTIS); 2019-002039-27 (EudraCT Number)
Record Dates: First submitted 2019-11-20; First posted 2019-12-09 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Hypereosinophilic Syndrome
Keywords: benralizumab; Hypereosinophilic Syndrome (HES)
MeSH Terms: conditions — Hypereosinophilic Syndrome | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All eligible patients will be centrally randomly assigned in a 1:1 ratio to receive either benralizumab or placebo. Randomisation will be done using an IWRS/IVRS.
  Benralizumab and placebo will not be visually distinct from each other. All packaging and labelling of the IP will be done in such a way as to ensure blinding for all Sponsor and investigational site staff. Neither the patient nor any of the Investigators or Sponsor staff who are involved in the treatment, clinical evaluation, and monitoring of the patients will be aware of the treatment received. Since benralizumab and placebo are not visually distinct, IP will be handled by an appropriately qualified member of the study team (e.g., pharmacist, Investigator, or designee) at the site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benralizumab arm (Experimental): 1x Benralizumab SC injection
  Interventions: Biological: Benralizumab
- Placebo arm (Placebo Comparator): 1x Benralizumab matching placebo SC injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Benralizumab — Benralizumab solution for injection in an accessorised prefilled syringe (APFS) will be administered subcutaneously (SC) every 4 weeks
  Arms: Benralizumab arm
Biological: Placebo — Matching placebo solution for injection in an APFS will be administered SC every 4 weeks
  Arms: Placebo arm

SUMMARY:
This is a multicentre, randomised, double-blind (DB), parallel-group, placebo-controlled, 24-week Phase III study to compare the efficacy and safety of benralizumab versus placebo administered by SC injection Q4W in patients with hypereosinophilic syndrome (HES). This study comprises 2 distinct periods (together defined as the 'main study'): A 24-week, DB treatment period, during which patients will be randomised to receive either benralizumab or placebo, in addition to their prior stable HES background therapy, and an open-label extension (OLE) period, during which all patients will receive benralizumab.

The primary database lock (DBL) will occur when approximately 38 patients have had their first HES worsening/flare event during the DB treatment period and all randomised patients have had the opportunity to be followed up for the 24-week DB treatment period.

A patient must complete the 24-week DB treatment period on investigational product (IP) to be eligible to enter the OLE treatment period. The final DBL will occur after the last patient completes the OLE.

DETAILED DESCRIPTION:
This is a multicentre, randomised, DB, parallel-group, placebo-controlled, 24-week Phase III study to compare the efficacy and safety of benralizumab 30 mg versus placebo administered by SC injection Q4W in patients with HES. This study will be conducted at approximately 68 sites in 18 countries.

The target patient population is male and female patients 12 years of age and older with symptomatic active HES. Eligible patients must be negative for the FIP1L1-PDGFRA fusion tyrosine kinase gene translocation.

Potentially eligible patients will enter a 3-day screening period and will be required to have documented stable HES therapy for at least 4 weeks prior to Visit 1 and AEC ≥ 1000 cells/μL at local laboratory testing to proceed to the second day of the screening period. Patients will be assessed for corticosteroid responsiveness (defined as an AEC < 1000 cells/μL after 2 days of OCS [prednisone/prednisolone] 1 mg/kg/day given on top of the patient's background therapy for HES) prior to randomisation; other OCSs in equivalent doses are permitted. Patients who are not corticosteroid responsive or fail any other eligibility criteria will be screen failed.

It is expected that approximately 120 patients will be randomised at a 1:1 ratio at the randomisation/baseline visit (Visit 3) to receive either benralizumab or matching placeboQ4W for a 24-week DB treatment period. Recruitment may continue beyond 120 patients if required to achieve the target number of HES worsening/flares. Recruitment of adolescent patients is targeted to be broadly in line with expected prevalence rates of adolescents in the overall population. Approximately 4 to 6 adolescent patients (aged 12 to 17) are targeted to be randomised. Randomisation will be stratified. Approximately 40 patients will participate in a noninterventional interview to collect data on HRQoL and the patients' experience during the DB portion of the study.

All patients will remain on stable dose(s) and regimen of background HES therapy during the screening period and throughout 36 weeks of treatment (until Visit 12/Week 36 when the therapy can be adjusted). During this time, background HES therapy may only be modified if a patient has an HES clinical worsening/flare or an AE thought to be due to background therapy.

AstraZeneca, sites, and patients will be blinded to the absolute eosinophil, basophil, and monocyte counts, differential blood counts (percentages) for all WBCs (eosinophils, basophils, monocytes, neutrophils, and lymphocytes), and biopsy cell counts (if applicable) after randomisation/baseline (Visit 3/Week 0), during the entire DB treatment period, and for the first 4 weeks of the OLE treatment period (until Visit 10/Week 28) after which no blinding to WBC counts or biopsy cell counts is required. After the primary DBL, AstraZeneca will become unblinded to all patients' blood and biopsy cell counts obtained during DB treatment period.

The final dose of the DB treatment period will be given at Week 20, and the DB treatment period will complete at Week 24.

All patients who complete the DB treatment period on IP may be eligible to continue into an OLE treatment period on benralizumab (30 mg SC Q4W). The OLE is intended to allow treatment with open-label benralizumab for at least 1 year for adults and at least 2 years for adolescents after completion of the DB treatment period of the study (earlier enrolled patients may therefore be in the OLE for longer than 1 year). AstraZeneca may choose to extend the study depending on the overall development program. Moreover, AstraZeneca reserves the right of terminating the OLE early (eg, if development of the asset is terminated or marketing authorisation is obtained).

The primary DBL will occur when approximately 38 patients have had their first HES worsening/flare event during the DB treatment period and all randomised patients have had the opportunity to be followed up for the 24-week DB treatment period. Treatment allocation will remain blinded until the primary DBL. A patient must complete the 24-week DB treatment period on IP to be eligible to enter the OLE treatment period. The final DBL will occur after the last patient completes the OLE. Data from the OLE treatment period of the study will be presented in an addendum to the primary analysis CSR and/or a separate OLE treatment period CSR.

ELIGIBILITY:
Inclusion Criteria

1. Provision of the signed and dated written informed consent of the patient or the patient's legally authorised representative, and informed assent from the patient (per local regulations) prior to any mandatory study-specific procedures, sampling, and analyses
2. Males and females 12 years of age and older at the time of signing the ICF
3. Documented diagnosis of HES (history of persistent eosinophilia > 1500 cells/μL without secondary cause on 2 examinations [interval ≥ 1 month; Valent et al 2012] and evidence of end organ manifestations attributable to the eosinophilia)
4. Documented negative testing for the FIP1L1-PDGFRA fusion tyrosine kinase gene translocation
5. Stable HES treatment dose(s) and regimen for ≥ 4 weeks at the time of Visit 1
6. Signs or symptoms of HES worsening/flare and/or laboratory abnormalities indicative of HES worsening/flare (other than isolated eosinophilia) at Visit 1 OR a documented history of 2 or more HES worsening/flares within 12 months prior to Visit 1 requiring an escalation in therapy

   a. At least one flare within the past 12 months must not be related to a decrease in HES therapy during the 4 weeks prior to the flare
7. AEC ≥ 1000 cells/μL at Visit 1 (assessed by local laboratory)
8. Corticosteroid responsiveness defined as an AEC < 1000 cells/μL after a 2-day course of OCS (prednisone/prednisolone) 1 mg/kg/day at Visit 2 (assessed by local laboratory). Other OCSs in equivalent doses are permitted
9. WOCBP must agree to use a highly effective method of birth control (confirmed by the investigator) from enrolment, throughout the study duration, and within 12 weeks after last dose of IP and have a negative urine dipstick pregnancy test result on Visit 1. Highly effective methods of birth control (those that can achieve a failure rate of less than 1% per year when used consistently and correctly) include:

   1. Combined (oestrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, or transdermal
   2. Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, or implantable
   3. Intrauterine device
   4. Intrauterine hormone-releasing system
   5. Bilateral tubal occlusion
   6. Sexual abstinence, ie, refraining from heterosexual intercourse (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient)
   7. Vasectomised sexual partner (provided that partner is the sole sexual partner of the WOCBP study patient and that the vasectomised partner has received medical assessment of the surgical success)

Exclusion Criteria

1. Life-threatening HES and/or HES complication(s) as judged by the investigator:

   1. Medical intervention for HES-related life-threatening event(s) within 12 weeks prior to randomization
   2. History of thrombotic complications, stroke, or significant cardiac damage related to HES, if the respective events were life threatening and currently represent a risk of life-threatening disease complications. Events that occurred in the past but considered resolved or stable, can be accepted if, as per investigator's judgment, participation in the study will not put the patient at risk
   3. Disease severity that in the opinion of the investigator makes the patient inappropriate for inclusion in the study
2. Presence of FIP1L1-PDGFRA fusion tyrosine kinase gene translocation or other known imatinib-sensitive mutation
3. Definitive diagnosis of eosinophilic granulomatosis with polyangiitis
4. Known, preexisting, clinically significant endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, haematological, respiratory, or any other system abnormalities that are not associated with HES and are uncontrolled with standard treatment which, in the opinion of the investigator, may put the patient at risk because of his/her participation in the study, or may influence the results of the study, or the patient's ability to complete the entire duration of the study
5. Hypereosinophilia of unknown significance
6. Cardiovascular: Documented history of any clinically significant cardiac damage, clinically significant echocardiography (if available) or ECG findings within 12 months prior to Visit 1 or clinically significant ECG findings at screening that in the opinion of the investigator may put the patients at risk
7. Known currently active liver disease

   1. Chronic stable hepatitis B and C (including positive testing for hepatitis B surface antigen or hepatitis C antibody) or other stable chronic liver disease are acceptable if patient otherwise meets eligibility criteria. Stable chronic liver disease should generally be defined by the absence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, oesophageal or gastric varices, or persistent jaundice, or cirrhosis
   2. ALT or AST level ≥ 3 × ULN during the screening period (AST or ALT > 5 × ULN if documented HES with liver manifestations). Transient increase of AST/ALT level that resolves by the time of randomisation is acceptable if, in the investigator's opinion, the patient does not have an active liver disease and meets other eligibility criteria
8. Current or history of malignancy within 5 years before the screening visit with the following exceptions:

   1. Patients treated for in situ carcinoma of the cervix who have completed curative therapy and are in remission for at least 12 months prior to signing the informed consent and
   2. Patients with basal cell or superficial squamous skin cancer
   3. Patients who have had other malignancies are eligible provided that the patient is in remission and curative therapy was completed at least 5 years prior to the date informed consent was obtained
9. Diagnosis of systemic mastocytosis
10. Chronic or ongoing active infections requiring systemic treatment, as well as clinically significant viral, bacterial, or fungal infection within 4 weeks prior to Visit 1
11. A helminth parasitic infection diagnosed within 24 weeks prior to Visit 1 that has not been treated or has failed to respond to standard of care therapy. A confirmation of a complete resolution of any helminth parasitic infection prior to Visit 1 should be available
12. A history of known immunodeficiency disorder other than that explained by the use of OCS or other therapy taken for HES. Positive HIV test

14. Evidence of prior benralizumab treatment failure

Ages: 12 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to first HES worsening/flare | Up to 24 weeks
  An HES worsening or flare is defined as HES clinical manifestations or lab abnormalities that result in an increase/burst of OCS ≥10 mg/day for at least 2 days, OR an increase or addition of new cytotoxic and/or immunosuppressive therapy, OR hospitalisation

SECONDARY OUTCOMES:
Proportion of patients who experience HES worsening/flare | Up to 24 weeks
  An HES worsening or flare is defined as HES clinical manifestations or lab abnormalities that result in an increase/burst of OCS ≥10 mg/day for at least 2 days, OR an increase or addition of new cytotoxic and/or immunosuppressive therapy, OR hospitalisation. For this endpoint patients who withdraw from the study without having flared are included in the analysis as a flare event.
number of HES worsenings/flares | Up to 24 weeks
  Number of HES worsenings/flares (annualised rate/year) during the DB period
Time to first haematologic relapse | Up to 24 weeks
  A haematologic relapse is defined as AEC ≥1000 cells/μL
Change from baseline in fatigue severity | at week 24
  Patient reported measure of fatigue severity (PROMIS fatigue short form 7a)
Proportion of patients who have haematologic relapse | Up to 24 weeks
  Proportion of patients who have haematologic relapse during the DB treatment period. Haematologic relapse post-baseline: AEC ≥ 1000 cells/μL. Patients who withdraw without having had a hematologic relapse will be considered as a relapse event in this analysis
Proportion of patients who have AEC<500 cells/µL for 24 weeks | Up to 24 weeks
  Proportion of patients who have AEC < 500 cells/μL for 24 weeks.
Proportion of patients who require an increase in corticosteroid dose | Up to 24 weeks
  Proportion of patients who require an increase in corticosteroid dose from baseline at any point in the double-blind treatment period
HRQoL | Up to 24 weeks
  Derived from the SF-36v2 questionnaires which contains 36 questions measuring patients' general functional health and well-being, both physically and mentally
PGIS | Up to 24 weeks
  The PGIS is a single question evaluating patients' perception of overall symptom severity
PGIC | Up to 24 weeks
  The PGIC is a single question evaluating whether there has been an improvement or decline in patients' overall health status after start of treatment.
Serum benralizumab concentration as a measure of pharmacokinetics | Up to 24 weeks
  Serum Benralizumab concentrations.
Anti-drug antibodies (ADA) titers and neutralizing antibodies (nAb) as measure of immunogenicity | Up to 24 weeks
  Anti-benralizumab antibodies and nAbs.
Adverse Events (AEs), vital signs and clinical laboratory assessments as an evaluation of safety and tolerability of benralizumab | Up to 24 weeks
  AEs, vital signs and clinical laboratory assessments.

CONTACTS AND LOCATIONS:
Locations (51):
- United States (8):
  - Research Site, La Jolla, California
  - Research Site, Atlanta, Georgia
  - Research Site, Bethesda, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Durham, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Salt Lake City, Utah
- Research Site, Rosario, Argentina
- Research Site, Innsbruck, Austria
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Edegem
- China (4):
  - Research Site, Chengdu
  - Research Site, Tianjin
  - Research Site, Xiamen
  - Research Site, Zhengzhou
- Research Site, København Ø, Denmark
- France (5):
  - Research Site, Lille
  - Research Site, Pessac
  - Research Site, Strasbourg
  - Research Site, Suresnes
  - Research Site, Toulouse
- Germany (3):
  - Research Site, Hanover
  - Research Site, Kirchheim
  - Research Site, Mannheim
- India (3):
  - Research Site, Ahmedabad
  - Research Site, Ajmer
  - Research Site, Delhi
- Israel (8):
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Rehovot
  - Research Site, Tel Aviv
- Research Site, Bologna, Italy
- Japan (7):
  - Research Site, Chiba
  - Research Site, Hamamatsu
  - Research Site, Ichikawa-shi
  - Research Site, Kawasaki-shi
  - Research Site, Nishinomiya-shi
  - Research Site, Osaka
  - Research Site, Sendai
- Research Site, Rotterdam, Netherlands
- Poland (3):
  - Research Site, Chęciny
  - Research Site, Gdansk
  - Research Site, Lodz
- Research Site, Seoul, South Korea
- Research Site, Santander, Spain
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home